CLINICAL TRIAL: NCT04290494
Title: Temporal Trends of Thrombolysis Treatment in Chinese Acute Ischemic Stroke (AIS) Patients From 2007 2017: Analysis of China National Stroke Registry (CNSR) I, II, and III
Brief Title: Temporal Trends of Thrombolysis Treatment in Chinese Acute Ischemic Stroke (AIS) Patients From 2007-2017: Analysis of China National Stroke Registry (CNSR) I, II, and III; CTP-Draft Review Performed;
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 0135-0343
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Results first posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CNSR I (2007 to 2008): For this group following patients will be analysed:
  The overall AIS patients aged 18 to 80 years who arrived at hospital within 7 days of symptom onset (Patient group A)
  Thereof: IVT eligible patients:
  AIS patients who arrived at hospital within 2 hours (patient group B) and 3.5 hours (patient group B') of symptom onset and with no documented absolute contraindications to IVT treatment
  Thereof: IV rtPA treated patients:
  IVT eligible patients who arrived at hospital within 2 hours of symptom onset and received IV rtPA within 3 hours of symptom onset (patient group C) and those who arrived at hospital within 3.5 hours of symptom onset and received IV rtPA within 4.5 hours of symptom onset (patient group C')
  Interventions: Drug: IV rtPA (intravenous recombinant plasminogen activator)
- CNSR II (2012 to 2013): For this group following patients will be analysed:
  The overall AIS patients aged 18 to 80 years who arrived at hospital within 7 days of symptom onset (Patient group A)
  Thereof: IVT eligible patients:
  AIS patients who arrived at hospital within 2 hours (patient group B) and 3.5 hours (patient group B') of symptom onset and with no documented absolute contraindications to IVT treatment
  Thereof: IV rtPA treated patients:
  IVT eligible patients who arrived at hospital within 2 hours of symptom onset and received IV rtPA within 3 hours of symptom onset (patient group C) and those who arrived at hospital within 3.5 hours of symptom onset and received IV rtPA within 4.5 hours of symptom onset (patient group C')
  Interventions: Drug: IV rtPA (intravenous recombinant plasminogen activator)
- CNSR III (2015 to 2017): For this group following patients will be analysed:
  The overall AIS patients aged 18 to 80 years who arrived at hospital within 7 days of symptom onset (Patient group A)
  Thereof: IVT eligible patients:
  AIS patients who arrived at hospital within 2 hours (patient group B) and 3.5 hours (patient group B') of symptom onset and with no documented absolute contraindications to IVT treatment
  Thereof: IV rtPA treated patients:
  IVT eligible patients who arrived at hospital within 2 hours of symptom onset and received IV rtPA within 3 hours of symptom onset (patient group C) and those who arrived at hospital within 3.5 hours of symptom onset and received IV rtPA within 4.5 hours of symptom onset (patient group C')
  Interventions: Drug: IV rtPA (intravenous recombinant plasminogen activator)

INTERVENTIONS:
Drug: IV rtPA (intravenous recombinant plasminogen activator) — intravenous injection

SUMMARY:
The present study is to be conducted based on the AIS patient data collected from CNSR I, II, and III.

The primary objectives are:

* To investigate the temporal changes in the proportion of intravenous recombinant plasminogen activator (IV rtPA) treatment from 2007 to 2017 among Intravenous Thrombolytics (IVT) eligible patients (patient groups B and B') and overall AIS patients (patient group A) in China;
* To investigate the temporal changes in IV rtPA treatment time intervals from 2007 to 2017 among IV rtPA treated patients (patient groups C and C') in China.

The secondary objectives are:

- To describe the demographic and clinical characteristics of the IV rtPA treated patients (patient groups C and C'), IVT eligible patients (patient groups B and B') and the overall AIS patients (patient group A) from 2007 to 2017 from the CNSR I to III.

ELIGIBILITY:
Inclusion Criteria:

* Patient group A: All AIS patients

  * Aged 18 80 years
  * Diagnosed with AIS on admission
* Patient groups B and B': IVT eligible patients

  * Met the in- and exclusion criteria of "all AIS patients"
  * Arrived at hospital within 2 h (patient group B) or 3.5 h (patient group B') of symptom onset
* Patient groups C and C': IV rtPA treated patients

  * Met the in- and exclusion criteria of "IVT eligible patients"
  * Treated with IV rtPA within 3 h (patient group C) or 4.5 h (patient group C') of symptom onset

Exclusion Criteria:

* Patient group A: All AIS patients

  * Missing baseline data including age and gender
  * Diagnosed with intracranial hemorrhage (ICH), Transient Ischemic Attack (TIA), subarachnoid hemorrhage (SAH), or unspecific stroke
  * Arrived at hospital after 7 days of symptom onset
* Patient groups B and B': IVT eligible patients

  * Missing key data including:

    i. symptom onset time (or last known well time) ii. hospital arrival time iii. whether received IVT treatment or not iv. the time of IVT treatment
  * Documented IVT absolute contraindications, according to the case report form (CRF) for each wave of CNSR
* Patient groups C and C': IV rtPA treated patients

  * Not received IVT
  * Received IVT other than rtPA
  * Treated with IV rtPA after 3 h (patient group C) or 4.5 h (patient group C') of symptom onset
  * Received additional treatments with intra arterial reperfusion or experimental therapies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible patients from the CNSR I to III will be included. Patient groups include the overall AIS patients (patient group A), IVT eligible patients (patient groups B and B'), and IV rtPA treated patients (patient groups C and C').
Sampling Method: Probability Sample
Enrollment: 42188 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://trials.boehringer-ingelheim.com/trial_results/clinical_submission_documents.html to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link http://trials.boehringer-ingelheim.com/ to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://trials.boehringer-ingelheim.com

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This non-interventional study was based on Chinese acute ischemic stroke patients who had treatment from 2007 to 2017 from the existing data of the China National Stroke Registry (CNSR) I, II, and III to investigate the temporal trends of thrombolysis treatment in Chinese acute ischemic stroke patients.
Pre-assignment Details: All eligible patients who met all inclusion and none of the exclusion criteria from the existing data of China National Stroke Registry (CNSR) I, II, and III with treatment from 2007 to 2017 were included.
Groups:
- China National Stroke Registry (CNSR) I (2007 to 2008): All eligible patients who met all inclusion and none of the exclusion criteria from the existing data of China National Stroke Registry (CNSR) I (data in this existing database were collected during 2007-2008) were included in this group.
- China National Stroke Registry (CNSR) II (2012 to 2013): All eligible patients who met all inclusion and none of the exclusion criteria from the existing data of China National Stroke Registry (CNSR) II (data in this existing database were collected during 2012-2013) were included in this group.
- China National Stroke Registry (CNSR) III (2015 to 2017): All eligible patients who met all inclusion and none of the exclusion criteria from the existing data of China National Stroke Registry (CNSR) III (data in this existing database were collected during 2015-2017) were included in this group.
Period: Overall Study
Arm/Group | China National Stroke Registry (CNSR) I (2007 to 2008) | China National Stroke Registry (CNSR) II (2012 to 2013) | China National Stroke Registry (CNSR) III (2015 to 2017)
Started | 10968 | 17823 | 13397
Completed | 10968 | 17823 | 13397
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All eligible patients who met all inclusion and none of the exclusion criteria from the existing data of China National Stroke Registry (CNSR) phase I to phase III with treatment from 2007 to 2017.
Groups:
- Total: Total of all reporting groups
Arm/Group | China National Stroke Registry (CNSR) I (2007 to 2008) | China National Stroke Registry (CNSR) II (2012 to 2013) | China National Stroke Registry (CNSR) III (2015 to 2017) | Total
Number analyzed (Participants) | 10968 | 17823 | 13397 | 42188
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.5 (11.1) | 62.9 (10.8) | 61.2 (10.4) | 62.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4053 | 6350 | 4114 | 14517
  Male | 6915 | 11473 | 9283 | 27671
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Received Intravenous Recombinant Plasminogen Activator (IV-rtPA) Treatment Within 3 Hours of Symptom Onset Among 2 Hours Intravenous Thrombolytics (IVT) Eligible Patients
Description: The percentage of patients who received Intravenous Recombinant Plasminogen Activator (IV-rtPA) treatment within 3 hours of symptom onset among patients eligible for intravenous thrombolytics (IVT) who arrived at the hospital within 2 hours since symptom onset was reported.
Time Frame: From 2007 to 2017, up to 10 years before this study started.
Population: All eligible patients who met all inclusion and none of the exclusion criteria from the existing data of China National Stroke Registry (CNSR) phase I to phase III with treatment from 2007 to 2017. Only those patients eligible for intravenous thrombolytics (IVT) who arrived at the hospital within 2 hours since symptom onset were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | China National Stroke Registry (CNSR) I (2007 to 2008) | China National Stroke Registry (CNSR) II (2012 to 2013) | China National Stroke Registry (CNSR) III (2015 to 2017)
Number analyzed (Participants) | 866 | 2214 | 1679
Percentage of participants | 11.66 [9.53 to 13.80] | 10.66 [9.37 to 11.94] | 28.77 [26.60 to 30.93]

2. Primary Outcome: Percentage of Patients Who Received Intravenous Recombinant Plasminogen Activator (IV-rtPA) Treatment Within 4.5 Hours of Symptom Onset Among 3.5 Hours Intravenous Thrombolytics (IVT) Eligible Patients
Description: The percentage of patients who received Intravenous Recombinant Plasminogen Activator (IV-rtPA) treatment within 4.5 hours of symptom onset among patients eligible for intravenous thrombolytics (IVT) who arrived at the hospital within 3.5 hours since symptom onset was reported.
Time Frame: From 2007 to 2017, up to 10 years before this study started.
Population: All eligible patients who met all inclusion and none of the exclusion criteria from the existing data of China National Stroke Registry (CNSR) phase I to phase III with treatment from 2007 to 2017. Only those patients eligible for intravenous thrombolytics (IVT) who arrived at the hospital within 3.5 hours since symptom onset were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | China National Stroke Registry (CNSR) I (2007 to 2008) | China National Stroke Registry (CNSR) II (2012 to 2013) | China National Stroke Registry (CNSR) III (2015 to 2017)
Number analyzed (Participants) | 1271 | 3684 | 2787
Percentage of participants | 13.53 [11.65 to 15.41] | 7.11 [6.28 to 7.94] | 33.44 [31.69 to 35.19]

3. Secondary Outcome: Percentage of Patients Who Arrived at Hospital Within 2 Hours of Symptom Onset and Who Received Intravenous Recombinant Plasminogen Activator (IV-rtPA) Treatment Within 3 Hours of Symptom Onset Among All Eligible Patients
Description: Percentage of patients who arrived at hospital within 2 hours of symptom onset and who received Intravenous Recombinant Plasminogen Activator (IV-rtPA) treatment within 3 hours of symptom onset among all eligible patients was reported.
Time Frame: From 2007 to 2017, up to 10 years before this study started.
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | China National Stroke Registry (CNSR) I (2007 to 2008) | China National Stroke Registry (CNSR) II (2012 to 2013) | China National Stroke Registry (CNSR) III (2015 to 2017)
Number analyzed (Participants) | 10968 | 17823 | 13397
Percentage of participants | 0.92 [0.74 to 1.10] | 1.32 [1.16 to 1.49] | 3.61 [3.29 to 3.92]

4. Secondary Outcome: Percentage of Patients Who Arrived at Hospital Within 3.5 Hours of Symptom Onset and Who Received Intravenous Recombinant Plasminogen Activator (IV-rtPA) Treatment Within 4.5 Hours of Symptom Onset Among All Eligible Patients
Description: Percentage of patients who arrived at hospital within 3.5 hours of symptom onset and who received Intravenous Recombinant Plasminogen Activator (IV-rtPA) treatment within 4.5 hours of symptom onset among all eligible patients was reported.
Time Frame: From 2007 to 2017, up to 10 years before this study started.
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | China National Stroke Registry (CNSR) I (2007 to 2008) | China National Stroke Registry (CNSR) II (2012 to 2013) | China National Stroke Registry (CNSR) III (2015 to 2017)
Number analyzed (Participants) | 10968 | 17823 | 13397
Percentage of participants | 1.57 [1.34 to 1.80] | 1.47 [1.29 to 1.65] | 6.96 [6.53 to 7.39]

5. Secondary Outcome: The Door to Needle (DTN) Time (Time Between Arrival at Hospital and the Administration of Intravenous Recombinant Plasminogen Activator (IV-rtPA) Treatment) Among 3 Hours IV-rtPA Treated Patients
Description: The door to needle (DTN) time (time between arrival at hospital and the administration of Intravenous Recombinant Plasminogen Activator (IV-rtPA) treatment) among patients who were treated with Intravenous Recombinant Plasminogen Activator (IV-rtPA) within 3 hours since symptom onset was reported.
Time Frame: From arrival at the hospital until the administration of Intravenous Recombinant Plasminogen Activator, up to 170 minutes.
Population: All eligible patients who met all inclusion and none of the exclusion criteria from the existing data of China National Stroke Registry (CNSR) phase I to phase III with treatment from 2007 to 2017. Only those patients who were treated with Intravenous Recombinant Plasminogen Activator (IV-rtPA) within 3 hours since symptom onset were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | China National Stroke Registry (CNSR) I (2007 to 2008) | China National Stroke Registry (CNSR) II (2012 to 2013) | China National Stroke Registry (CNSR) III (2015 to 2017)
Number analyzed (Participants) | 101 | 236 | 483
minutes | 90.0 [60.0 to 120.0] | 100.0 [74.0 to 113.0] | 58.0 [38.0 to 77.0]

6. Secondary Outcome: Percentage of Patients With Door to Needle (DTN) Time (Time Between Arrival at Hospital and the Administration of Intravenous Recombinant Plasminogen Activator (IV-rtPA) Treatment) ≤ 60 Minutes Among 3 Hours IV-rtPA Treated Patients
Description: The percentage of patients with door to needle (DTN) time (time between arrival at hospital and the administration of Intravenous Recombinant Plasminogen Activator (IV-rtPA) treatment) ≤ 60 minutes among patients who were treated with Intravenous Recombinant Plasminogen Activator (IV-rtPA) within 3 hours since symptom onset was reported.
Time Frame: From 2007 to 2017, up to 10 years before this study started.
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | China National Stroke Registry (CNSR) I (2007 to 2008) | China National Stroke Registry (CNSR) II (2012 to 2013) | China National Stroke Registry (CNSR) III (2015 to 2017)
Number analyzed (Participants) | 101 | 236 | 483
Percentage of participants | 28.71 [19.89 to 37.54] | 12.29 [8.1 to 16.48] | 59.21 [54.83 to 63.6]

7. Secondary Outcome: Time Between Symptom Onset and Arrival at Hospital Among 3 Hours Intravenous Recombinant Plasminogen Activator (IV-rtPA) Treated Patients
Description: Time between symptom onset and arrival at hospital among patients who were treated with Intravenous Recombinant Plasminogen Activator (IV-rtPA) within 3 hours since symptom onset was reported.
Time Frame: From symptom onset until arrival at the hospital, up to 120 minutes.
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | China National Stroke Registry (CNSR) I (2007 to 2008) | China National Stroke Registry (CNSR) II (2012 to 2013) | China National Stroke Registry (CNSR) III (2015 to 2017)
Number analyzed (Participants) | 101 | 236 | 483
minutes | 60.0 [32.0 to 90.0] | 59.0 [43.0 to 75.0] | 69.0 [50.0 to 93.0]

8. Secondary Outcome: Time Between Symptom Onset and the Administration of Intravenous Recombinant Plasminogen Activator (IV-rtPA) Treatment Among 3 Hours IV-rtPA Treated Patients
Description: Time between symptom onset and the administration of Intravenous Recombinant Plasminogen Activator (IV-rtPA) treatment among patients who were treated with Intravenous Recombinant Plasminogen Activator (IV-rtPA) within 3 hours since symptom onset was reported.
Time Frame: From symptom onset until administration of Intravenous Recombinant Plasminogen Activator, up to 180 minutes.
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | China National Stroke Registry (CNSR) I (2007 to 2008) | China National Stroke Registry (CNSR) II (2012 to 2013) | China National Stroke Registry (CNSR) III (2015 to 2017)
Number analyzed (Participants) | 101 | 236 | 483
minutes | 150.0 [138.0 to 170.0] | 156.0 [141.0 to 165.0] | 134.0 [108.0 to 155.0]

9. Secondary Outcome: The Door to Needle (DTN) Time (Time Between Arrival at Hospital and the Administration of Intravenous Recombinant Plasminogen Activator (IV-rtPA) Treatment) Among 4.5 Hours IV-rtPA Treated Patients
Description: The door to needle (DTN) time (time between arrival at hospital and the administration of Intravenous Recombinant Plasminogen Activator (IV-rtPA) treatment) among patients who were treated with Intravenous Recombinant Plasminogen Activator (IV-rtPA) within 4.5 hours since symptom onset was reported.
Time Frame: From arrival at the hospital until the administration of Intravenous Recombinant Plasminogen Activator, up to 247 minutes.
Population: All eligible patients who met all inclusion and none of the exclusion criteria from the existing data of China National Stroke Registry (CNSR) phase I to phase III with treatment from 2007 to 2017. Only those patients who were treated with Intravenous Recombinant Plasminogen Activator (IV-rtPA) within 4.5 hours since symptom onset were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | China National Stroke Registry (CNSR) I (2007 to 2008) | China National Stroke Registry (CNSR) II (2012 to 2013) | China National Stroke Registry (CNSR) III (2015 to 2017)
Number analyzed (Participants) | 172 | 262 | 932
minutes | 94.0 [60.0 to 130.0] | 95.0 [72.0 to 112.0] | 60.0 [38.0 to 84.5]

10. Secondary Outcome: Percentage of Patients With Door to Needle (DTN) Time (Time Between Arrival at Hospital and the Administration of Intravenous Recombinant Plasminogen Activator (IV-rtPA) Treatment) ≤ 60 Minutes Among 4.5 Hours IV-rtPA Treated Patients
Description: The percentage of patients with door to needle (DTN) time (time between arrival at hospital and the administration of Intravenous Recombinant Plasminogen Activator (IV-rtPA) treatment) ≤ 60 minutes among patients who were treated with Intravenous Recombinant Plasminogen Activator (IV-rtPA) within 4.5 hours since symptom onset was reported.
Time Frame: From 2007 to 2017, up to 10 years before this study started.
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | China National Stroke Registry (CNSR) I (2007 to 2008) | China National Stroke Registry (CNSR) II (2012 to 2013) | China National Stroke Registry (CNSR) III (2015 to 2017)
Number analyzed (Participants) | 172 | 262 | 932
Percentage of participants | 26.74 [20.13 to 33.36] | 13.36 [9.24 to 17.48] | 53.43 [50.23 to 56.64]

11. Secondary Outcome: Time Between Symptom Onset and Arrival at Hospital Among 4.5 Hours Intravenous Recombinant Plasminogen Activator (IV-rtPA) Treated Patients
Description: Time between symptom onset and arrival at hospital among patients who were treated with Intravenous Recombinant Plasminogen Activator (IV-rtPA) within 4.5 hours since symptom onset was reported
Time Frame: From symptom onset until arrival at the hospital, up to 210 minutes.
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | China National Stroke Registry (CNSR) I (2007 to 2008) | China National Stroke Registry (CNSR) II (2012 to 2013) | China National Stroke Registry (CNSR) III (2015 to 2017)
Number analyzed (Participants) | 172 | 262 | 932
minutes | 75.0 [42.5 to 110.0] | 59.0 [45.0 to 84.0] | 100.0 [60.0 to 140.0]

12. Secondary Outcome: Time Between Symptom Onset and the Administration of Intravenous Recombinant Plasminogen Activator (IV-rtPA) Treatment Among 4.5 Hours IV-rtPA Treated Patients
Description: Time between symptom onset and the administration of Intravenous Recombinant Plasminogen Activator (IV-rtPA) treatment among patients who were treated with Intravenous Recombinant Plasminogen Activator (IV-rtPA) within 4.5 hours since symptom onset was reported
Time Frame: From symptom onset until the administration of Intravenous Recombinant Plasminogen Activator, up to 270 minutes.
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | China National Stroke Registry (CNSR) I (2007 to 2008) | China National Stroke Registry (CNSR) II (2012 to 2013) | China National Stroke Registry (CNSR) III (2015 to 2017)
Number analyzed (Participants) | 172 | 262 | 983
minutes | 175.0 [150.0 to 200.0] | 159.0 [144.0 to 169.0] | 170.0 [132.0 to 210.0]

ADVERSE EVENTS:
Time Frame: Adverse event information was not collected for this study.
Description: As this was a non-interventional study with secondary use of existing data from China National Stroke Registry (CNSR) I, II, and III database, safety data were not collected and adverse events reporting on an individual case level is not applicable. The "0" in the Number Affected and Number At Risk in the All-Cause Mortality, Serious Adverse Event, and Other (non-serious) Adverse Events sections stands for mortality, serious and other (non-serious) adverse events were not collected.
Arm/Group | China National Stroke Registry (CNSR) I (2007 to 2008) | China National Stroke Registry (CNSR) II (2012 to 2013) | China National Stroke Registry (CNSR) III (2015 to 2017)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-04-17): https://cdn.clinicaltrials.gov/large-docs/94/NCT04290494/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/94/NCT04290494/SAP_001.pdf